CLINICAL TRIAL: NCT03770871
Title: Evaluation of Resin Modified Glass Ionomer Liner (Vitrebond™) Versus Calcium Hydroxide as Indirect Pulp Treatment Material Used in Deep Carious Lesions in Primary Molars: A Randomized Clinical Trial
Brief Title: Indirect Pulp Treatment in Primary Molars
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Rashed, Researcher assisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2014-11-3
Record Dates: First submitted 2018-08-18; First posted 2018-12-10 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Dental Caries
Keywords: indirect pulp; primary; calcium hydroxide; resin modified glass ionomer; Children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Parallel group with 1:1 allocation ratio
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IPT using Dycal (TM ) (Active Comparator): Indirect pulp treatment; IPT using Dycal (TM ); (2 paste system) by partial caries removal
  Interventions: Drug: Indirect pulp treatment using Dycal (TM); Drug: Indirect pulp treatment using Vitrebond (TM )
- IPT using Vitrebond (TM ) (Experimental): Indirect pulp treatment; IPT using Vitrebond (TM );(powder and liquid) by partial caries removal
  Interventions: Drug: Indirect pulp treatment using Dycal (TM); Drug: Indirect pulp treatment using Vitrebond (TM )

INTERVENTIONS:
Drug: Indirect pulp treatment using Dycal (TM) — Partial caries removal and protection of the dental pulp with biocompatible material
  Other Names: Indirect pulp capping
Drug: Indirect pulp treatment using Vitrebond (TM ) — Partial caries removal and protection of the dental pulp with biocompatible material
  Other Names: Indirect pulp capping

SUMMARY:
This study was conducted to evaluate the clinical and the radiographic success of Dycal and Vitrebond as indirect pulp treatment materials in primary molars.

DETAILED DESCRIPTION:
Evaluation of calcium hydroxide and resin modified glass ionomer liner clinically and radiographically as indirect pulp treatment materials in deep caries in primary molars.

ELIGIBILITY:
Inclusion criteria:

In compliance with AAPD, 2017 guidelines for pulp therapy "IPT is indicated in a primary tooth with no pulpitis or with reversible pulpitis when the deepest carious dentin is not removed to avoid a pulp exposure. The pulp is judged by clinical and radiographic criteria to be vital and able to heal from the carious insult"

In addition to:

I-Subjects:

1. Medically free children, their parent(s) accepts to sign the informed consent.
2. Age range from 4-8 years.

II-Molars:

1. Presence of at least 1 primary molar with deep carious lesion extending to more than one half of the dentin on radiographic examination (to make the trial regardless of number of carious molars).
2. Clinically: Normal mobility and normal appearance of gingiva (vital teeth).
3. Radiographically: Normal roots without physiological resorption, normal lamina dura and normal periodontal membrane space (indicated for IPT).

Exclusion criteria:

I-Subjects:

1. Uncooperative children.
2. Parents unable to attend follow up visits (even after explaining the importance of recall visits).

II-Molars:

1. History of spontaneous pain (to exclude reversible pulpitis).
2. Clinically: Presence of swelling, sinus, fistula or tooth mobility (to exclude non vital teeth).
3. Radiographically: Presence of radiolucent lesions at furcation or periapical region or external or internal resorption (to exclude teeth not indicated for IPT).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of cases reporting postoperative pain | 12 months
  Presence of postoperative pain following dental treatment through patient questionnaire as a sign of clinical failure
Number of cases reporting swelling | 12 months
  Presence of postoperative swelling following dental treatment through visual examination using hand mirror as a sign of clinical failure
Number of cases reporting sinus | 12 months
  Presence of sinus following dental treatment through visual examination using hand mirror as a sign of clinical failure
Number of cases reporting fistula | 12 months
  Presence of fistula following dental treatment through visual examination using hand mirror as a sign of clinical failure
Number of cases reporting tooth mobility | 12 months
  Presence of abnormal tooth mobility following dental treatment through tactile examination using two hand mirrors as a sign of clinical failure

SECONDARY OUTCOMES:
Number of cases reporting external root resorption | 12 months
  Occurrence of pathological external root resorption following dental treatment through parallel periapical radiographic examination as a sign of radiographic failure
Number of cases reporting internal root resorption | 12 months
  Occurrence of pathological internal root resorption following dental treatment through parallel periapical radiographic examination as a sign of radiographic failure
Number of cases reporting furcation involvement | 12 months
  Occurrence of pathological internal root resorption following dental treatment through parallel periapical radiographic examination as a sign of radiographic failure
Number of cases reporting widening of periodontal membrane space | 12 months
  Occurrence of widening of periodontal membrane space following dental treatment through parallel periapical radiographic examination as a sign of radiographic failure
Number of cases reporting periapical radiolucency | 12 months
  Occurrence of periapical radiolucency following dental treatment through parallel periapical radiographic examination as a sign of radiographic failure

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Taha, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
final results